CLINICAL TRIAL: NCT00403962
Title: A Randomised, Double-Blind, Parallel-Group, Placebo-Controlled Fixed Dose Study Comparing the Efficacy and Safety of GW597599/Paroxetine Combination or Paroxetine Monotherapy to Placebo in Patients With Social Anxiety Disorder (SAD)
Brief Title: A Combination Therapy In Patients With Social Anxiety Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NKP103401
Record Dates: First submitted 2005-08-29; First posted 2006-11-27 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Social Phobia
Keywords: anxiety; Social Anxiety Disorder; SAD
MeSH Terms: conditions — Phobia, Social; Anxiety Disorders | interventions — vestipitant; Paroxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: vestipitant/paroxetine

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of a combination of Vestipitant and Paroxetine in patients with Social Anxiety Disorder (SAD)

ELIGIBILITY:
Inclusion criteria:

* Primary diagnosis of Generalised Social Anxiety Disorder as defined in DSM-IV.
* Capable of giving informed consent and willing to comply with the study requirements.
* Women of childbearing potential must agree to one of a number of defined acceptable methods of birth control.

Exclusion criteria:

* Primary diagnosis within the past 6 months of another Axis 1 disorder such as Major Depression or another anxiety disorder.
* Use of medications for a psychiatric condition including herbals in the past 2-12 weeks according to medication type.
* Subjects who, in the investigator's judgement pose a current, serious suicidal or homicidal risk or have made a suicide attempt within the past 6 months.
* Subjects who currently meet or who met within 6 months prior to screening DSM-IV criteria for substance abuse or subjects who currently meet or who met within 6 months prior to screening DSM-IV criteria for substance dependence (other than nicotine).
* Significantly abnormal blood or urine laboratory tests or electrocardiogram (ECG).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 204
Dates: Start 2004-11; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Change in score on a Social Anxiety Disorder rating scale following 12 weeks of treatment.

SECONDARY OUTCOMES:
Change in score on a number of rating scales following 12 weeks of treatment assessing symptomatic, behavioural and functional parameters which together provide a more complete description of the disorder.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- Denmark (7):
  - GSK Investigational Site, Hilleroed
  - GSK Investigational Site, Hvidovre
  - GSK Investigational Site, Koebenhavn K
  - GSK Investigational Site, Koebenhavn OE
  - GSK Investigational Site, Risskov
  - GSK Investigational Site, Skanderborg
  - GSK Investigational Site, Soroe
- Germany (3):
  - GSK Investigational Site, Hüttenberg, Hesse
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Berlin, State of Berlin
- Norway (4):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Hamar
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Sandvika
- South Africa (2):
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Tygerberg

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: NKP103401 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: NKP103401 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: NKP103401 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: NKP103401 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: NKP103401 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: NKP103401 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: NKP103401 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register